CLINICAL TRIAL: NCT06006494
Title: Comparison of the Effectiveness of Yoga and Exercise in Female Patients With Fibromyalgia Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Dr. Öğr. Üyesi Ömer Şevgin, Asst.Prof.Dr., Uskudar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Uskudar53
Record Dates: First submitted 2023-08-17; First posted 2023-08-23 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Fibromyalgia
Keywords: women; sleep; tiredness
MeSH Terms: conditions — Fibromyalgia; Fatigue | interventions — Yoga

STUDY DESIGN:
Intervention Model Description: Aerobic exercises, resistant exercises and yoga
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- aerobic group (Active Comparator): only a separate aerobic exercise will be given
  Interventions: Other: aerobic
- resistant group (Experimental): aerobic and resistance exercises will be given
  Interventions: Other: aerobic; Other: resistant
- yoga group (Experimental): aerobic exercises will be given and yoga will be done
  Interventions: Other: aerobic; Other: yoga

INTERVENTIONS:
Other: aerobic — We can think of aerobic exercise as a low-intensity long-term activity using large muscle groups (between 60-80% of maximal heart rate). For example; includes activities such as walking, cycling, jogging, aerobic dancing, swimming.
  An average of 50 minutes of exercise per day will be required, 3 days a week.
Other: resistant — Resistance exercises are the whole of the exercises in which effort is made against the weight and the weight is lifted. Exercises with therabands, dumbbells or body weight will be given. The exercises will be done 2 days a week for an average of 30-40 minutes.
  Arms: resistant group
Other: yoga — Yoga is basically breathing exercises, warm-up exercises, relaxation, It is a session consisting of movements and relaxation exercises.movements are performed by standing in a fixed posture for 15 seconds to 2 minutes in a certain posture, they are postures for both strengthening, stretching and balance. Yoga practice will be done 2 days a week for an average of 40 minutes.
  Arms: yoga group

SUMMARY:
In this study, yoga, aerobic exercise, resistance exercise training in female individuals with fibromyalgia syndrome; It was aimed to compare their effectiveness on fatigue, quality of life and pain.

DETAILED DESCRIPTION:
The study was planned as a randomized controlled study. Participants will be divided into 3 groups by simple randomization method. groups will be named as aerobic, yoga and resistance exercise groups. 12-week exercise protocols will be applied to all participants. Participants before and after treatment; The Fibromyalgia Impact Questionnaire, the McGill Pain Questionnaire for pain assessment, the Chalder Fatigue Scale to assess their fatigue level, will be filled in by the participants before and after the study. The data obtained will be statistically analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-45
* Be woman
* Being diagnosed with fibromyalgia

Exclusion Criteria:

* Receiving pharmacological treatment
* Having had a surgical operation in the last 6 months
* Being pregnant
* Having a musculoskeletal injury

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-12-10 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Fibromyalgia Impact Questionnaire | 14 weeks
  It assesses the impact of fibromyalgia on the patient's health and functional abilities.
  High scores indicate that the disease affects the person more. The total score can be between 0-80. A score of 80 indicates high influence.

CONTACTS AND LOCATIONS:
Overall Officials: Hilal ATASOY, Study Chair — Uskudar University
Locations (1):
- Uskudar University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sosa-Reina MD, Nunez-Nagy S, Gallego-Izquierdo T, Pecos-Martin D, Monserrat J, Alvarez-Mon M. Effectiveness of Therapeutic Exercise in Fibromyalgia Syndrome: A Systematic Review and Meta-Analysis of Randomized Clinical Trials. Biomed Res Int. 2017;2017:2356346. doi: 10.1155/2017/2356346. Epub 2017 Sep 20. PMID 29291206
- [Background] Busch AJ, Webber SC, Brachaniec M, Bidonde J, Bello-Haas VD, Danyliw AD, Overend TJ, Richards RS, Sawant A, Schachter CL. Exercise therapy for fibromyalgia. Curr Pain Headache Rep. 2011 Oct;15(5):358-67. doi: 10.1007/s11916-011-0214-2. PMID 21725900
- [Background] Bidonde J, Busch AJ, Schachter CL, Overend TJ, Kim SY, Goes SM, Boden C, Foulds HJ. Aerobic exercise training for adults with fibromyalgia. Cochrane Database Syst Rev. 2017 Jun 21;6(6):CD012700. doi: 10.1002/14651858.CD012700. PMID 28636204
- [Background] Busch AJ, Webber SC, Richards RS, Bidonde J, Schachter CL, Schafer LA, Danyliw A, Sawant A, Dal Bello-Haas V, Rader T, Overend TJ. Resistance exercise training for fibromyalgia. Cochrane Database Syst Rev. 2013 Dec 20;2013(12):CD010884. doi: 10.1002/14651858.CD010884. PMID 24362925
- [Background] Verma A, Shete SU, Doddoli G. Yoga therapy for fibromyalgia syndrome: A case report. J Family Med Prim Care. 2020 Jan 28;9(1):435-438. doi: 10.4103/jfmpc.jfmpc_816_19. eCollection 2020 Jan. PMID 32110633
- [Derived] Sevgin O, Bugday B, Aydogan Baykara R, Gunendi G, Akkurt B, Atasoy H, Dikmen Hosbas B, Akkurt MF, Karamancioglu B. Efficacy of different exercises in women with fibromyalgia syndrome: a randomised controlled trial. Clin Exp Rheumatol. 2025 Jun;43(6):1010-1018. doi: 10.55563/clinexprheumatol/uol8so. Epub 2025 Feb 12. PMID 39946182